CLINICAL TRIAL: NCT01942460
Title: Use of FERAHEME® (Ferumoxytol) for Severe Chronic Kidney Disease and Peritoneal Dialysis
Brief Title: Ferumoxytol for Iron-Deficiency Anemia in Chronic Kidney Disease and Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Georges Ouellet (Other)
Responsible Party: Sponsor-Investigator, Georges Ouellet, Nephrologist, Maisonneuve-Rosemont Hospital
Organization: Maisonneuve-Rosemont Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FER-CA-IIT-001
Record Dates: First submitted 2013-09-06; First posted 2013-09-16 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Iron-Deficiency Anemia; Inflammation; Oxidative Stress
Keywords: Iron; Anemia; Chronic Kidney Disease; Peritoneal Dialysis; Inflammation; Oxidative stress
MeSH Terms: conditions — Anemia, Iron-Deficiency; Inflammation; Anemia; Renal Insufficiency, Chronic | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ferumoxytol (Experimental)
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol
  Other Names: Feraheme

SUMMARY:
The purpose of this study is to investigate the efficacy of ferumoxytol for the repletion of iron stores and correction of iron deficiency anaemia in patients with severe chronic kidney disease or end-stage chronic kidney disease on peritoneal dialysis, and to assess the impact of the administration of a ferumoxytol dose on various markers for iron stores, as well as on various markers for inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* For women of childbearing age, negative serum pregnancy test at screening.
* Severe chronic kidney disease (TFGe lower than 30 ml/min) OR end-stage kidney disease on peritoneal dialysis.
* Anaemia, as defined by haemoglobin (Hb) < 120 g/L, within 14 days prior to screening, in a patient with or without an Erythropoiesis-stimulating agent (ESA).
* Iron depletion, as defined by transferrin saturation (TSAT) < 20% and/or a ferritin assay (FERR) < 200, within 14 days prior to screening.
* If an ESA is used, stable dose over the past 60 days.

Exclusion Criteria:

* Allergy to ferumoxytol or another intravenous iron formulation.
* Administration of ferumoxytol or any other intravenous, intramuscular or oral iron formulation within 30 days of enrolment.
* Patient who have received a blood transfusion within 2 weeks prior to enrolment, or are planned to receive a blood transfusion over the duration of the study.
* Patient currently participating in a clinical trial with another investigational drug or device or who have received an investigational drug or device within 30 days of enrolment in this study.
* Hb < 90 g/L at the time of screening.
* Existing or clinically suspected bleeding of digestive, gynaecological or other origin.
* Patient who have another cause of anemia, other than iron deficiency (for example, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, multiple myeloma, myelodysplastic disorder, etc.).
* Patients who are not responding to ESA or who are receiving in excess of 30000 units/week of erythropoietin (EPO), or 150 mcg/week of darbepoietin alfa.
* Major surgery within one month prior to enrolment in the study or planned surgery, other than vascular access creation, while the patient is in on the study.
* Patient who have had a malignancy (except for non-melanoma cancer of the skin) unless the patient has received curative treatment and has been disease-free for > 2 years.
* Patient who are considered by the Investigator to have a medical status that would preclude the patient's participation in this protocol.
* Patient due to have a magnetic resonance imaging examination or in whom such an examination is planned, in the next three months.
* Woman who plans to become pregnant in the next three months.
* Woman that is breastfeeding.
* Ongoing or recent (< 2 weeks) bacterial infection requiring treatment.
* Patient unable to give informed consent.
* Patient refuses to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin, serum ferritin and transferrin saturation | 4 weeks following ferumoxytol administration

SECONDARY OUTCOMES:
Change in inflammatory markers (C-reactive protein and Interleukin-6) | 60 minutes following ferumoxytol administration
Change in oxidative stress markers (Malondialdehyde, Advance Oxidation Protein Products, Non Transferrin-bound Iron) | 60 minutes following ferumoxytol administration
Change in soluble transferrin receptor | 4 weeks following ferumoxytol administration

CONTACTS AND LOCATIONS:
Overall Officials: Georges Ouellet, MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada